CLINICAL TRIAL: NCT03169491
Title: Caliber of Upper Airway Measured by Acoustic Pharyngometry in Children With Obstructive Sleep Apnea Before and After the Use of Presurgical CPAP and After Adentonsillectomy, and Their Relation With Surgical Complications and Residual Apneas
Brief Title: Effect of CPAP and Adenotonsillectomy in Upper Airway Volume of Children With OSAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Angélica Margarita Portillo Vásquez, PhD Student, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C12-16
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2018-07

CONDITIONS: Sleep Apnea, Obstructive; Child; Continuous Positive Airway Pressure; Adenoidectomy; Tonsillectomy
Keywords: Sleep Apnea, Obstructive; Child; Continuous Positive Airway Pressure; Perioperative management; Adenotonsillectomy; Acoustic pharyngometry
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: All recruited children with diagnosis of mild to moderate OSAS will be randomized to suboptimal (CPAP at 4 cmH2O) or therapeutical (CPAP auto from 4 to 15 cmH2O) arms, from a predetermined list in two groups of 50, blocks of 10 patients. All patients with diagnosis of severe OSAS will receive therapeutic pressure, and are considered as part of a third arm not included in the sample size.
Who Masked: Participant, Investigator
Masking Description: The CPAP equipment will be programed by the technician, not knowing the children, the parents or the main researcher whether the pressure is suboptimal or therapeutic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Therapeutic (Experimental): Continuous positive airway pressure (CPAP) with automatic pressure from 4 to 15 cmH2O every night for one week, afterwards use of CPAP at the P90 of pressure determinated during automatic use for one week, via oronasal interface.
  Interventions: Device: Continuous positive airway pressure (CPAP)
- Suboptimal (Sham Comparator): Continuous positive airway pressure (CPAP) every night for two weeks at fixed pressure of 4 cmH2O, via oronasal interface.
  Interventions: Device: Continuous positive airway pressure (CPAP)
- Severe OSAS (Other): Continuous positive airway pressure (CPAP) with automatic pressure from 4 to 15 cmH2O every night for one week, afterwards use of CPAP at the P90 of pressure determinated during automatic use for one week, via oronasal interface.
  Interventions: Device: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — CPAP dispositives will be used by the children in the study every night for two weeks. Devices AutoSet Spirit from ResMed.

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) in children has high prevalence and severe complications, and its first line of treatment (adenotonsillectomy) has risk of complications. Even though the use of presurgical CPAP seems logical due to its effects in adults, it must be studied in children due to the different physiopathology and adherence. One non-invasive way of study the effect is via acoustic pharyngometry, which can measure the anatomical site of obstruction. The post-surgical anatomical changes could correlate with a persistent OSAS, which would be helpful in selecting those patients who require a post surgical sleep study. The main goal of the study is to cuantify the changes in the oropharyngeal volume via acoustic pahryngometry after CPAP use, and also the changes after adentonsillectomy in children.

DETAILED DESCRIPTION:
The obstructive sleep apnea syndrome (OSAS) is defined as recurrent events of obstruction of the upper airway (with alteration of normal oxygenation, ventilation or sleep pattern). In children originates complications such as cognitive, cardiovascular and metabolic disorders and growth failure, which make its management imperative. It has a reported prevalence between 1 and 5%, highest between 2 and 8 years old, due to tonsil and adenoid hypertrophy, which causes obstruction of the upper airway, unlike the fat deposits of adults. This physiopathological cause of obstruction makes adenotonsillectomy the first line of management. This is a secure procedure, which still has an incidence of complications of 19%, (9.5% respiratory and 2.4% secondary bleeding). Those with OSAS present complications more frequently than those without7. Even though the surgery is considered succesful, up to 21.6% of those treated present persistence of the disease. Based on these results the American Academy of Pediatrics recommends considering polysomnography after surgery in those patients with high risk of persistence, such as obese children.

The continuous positive airway pressure (CPAP) device provides a continuous pressure through a mask, acting as a pneumatic ferule which keeps the upper airway permeable; with a lower possibility of obstruction. The adherence of pediatric patients to CPAP has been reported between 6 and 65% (which is one of the reasons it's not considered the first line treatment), with an use of 2.1 to 8.2 hours per night, and an AIH (apnea-hypopnea index) between 2 and 6 per hour. In adult patients, a reduction in trans and post-surgical risk has been found, and therefore its pre-surgical use is recommended. In children it is one of the strategies used to reduce surgical risk in OSAS, even though its use is not recommended in any of the main clinical guides of management of children with OSAS. Its use has been described in children with severe illness, and in other studies it was used in 18% of patients, but its real effect in the probable complications has not been prospectively studied.

In adult subjects, inflammation of upper airway has been reported, and it could play a role in the physiopathology of OSAS, with changes in the minimal sectional area and pharyngeal volume measured by MRI after use for 4 to 6 weeks of CPAP use. Albeit the physiopathology is not completely understood, it could be a consequence of the mechanical stress associated to obstruction of airflow, with the repeated trauma related with snore, jointly with the upper airway vibration and the suction from the collapse during the apneas the causes. CPAP eliminates respiratory events, which could cause a reduction in edema and inflammation.

Acoustic pharyngometry is a non-invasive method which uses sound reflection to quickly measure the sectional area of the upper airway in function of the distance from the oral aperture. It can be adapted to its use in children, obtaining highly reproducible results, even though it is limited to those who can follow instructions. In adults a difference was found between the minimum oropharyngeal area and the mean area after 1 week of CPAP use, but not between 1 week and 6 months of use, with a return to basal after a 1 week of nonuse. In our center change in volume and transversal oropharyngeal area have been found with acoustic pharyngometry since the second week of use of CPAP, of 5% at 2 weeks and 6% at 4 weeks. In children changes after surgery have been found, with increase in the minimal sectional area and oropharyngeal volume, even though its correlation with persistent OSAS has not been studied.

In order to study the changes in the upper airway after CPAP, acoustic pharyngometry will be performed before and after CPAP use, and 3 months after adenotonsillectomy to determinate the relation to persistent OSAS. The presurgical CPAP will be randomized in those children with diagnosis of mild to moderate OSAS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4 and 14 years old. Both genders. Diagnosis of OSAS based on sleep study (respiratory polygraphy or polysomnography).

Surgical treatment planned by the ORL department of the Institute of Respiratory Diseases of Mexico.

Residents of the Metropolitan Area of Mexico City Parents and child accept to particpate in the study, singning informed consent and assent.

Exclusion Criteria:

* Previous surgery in upper airway. Craneofacial malformation. Previous use of CPAP. Syndromatic patient.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2016-07-04 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Oropharyngeal volume postCPAP. | After two weeks of CPAP use.
  Upper airway volume as measured by acoustic pharyngometry.

SECONDARY OUTCOMES:
Oropharyngeal volume post-surgery | Three months after adenotonsillectomy.
  Upper airway volume as measured by acoustic pharyngometry.
OSA-18. | After two weeks of CPAP use.
  Score in que quality of life questionnaire OSA-18.
OSA-18. | Three months after adenotonsillectomy.
  Score in que quality of life questionnaire OSA-18.
Pediatric Sleep Questionnaire. | After two weeks of CPAP use.
  Symptoms as described in the pediatric sleep questionnaire.
Pediatric Sleep Questionnaire. | Three months after adentonsillectomy.
  Symptoms as described in the pediatric sleep questionnaire.
Surgical complications. | During and one month after surgery.
  Complications during or after the surgical procedure, as determined by checklist.

OTHER OUTCOMES:
Residual respiratory disturbance index. | Three months after adenotonsillectomy.
  Number of events of apnea, hypopnea per hour as measured by type 3 sleep monitor.

CONTACTS AND LOCATIONS:
Overall Officials: José Rogelio Pérez-Padilla, MD, Study Director — Instituto Nacional Enfermedades Respiratorias
Locations (1):
- Instituto Nacional Enfermedades Respiratorias, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Data from the study could be provided if solicited at the main author's e-mail adress.

REFERENCES:
- [Background] Kaditis AG, Alonso Alvarez ML, Boudewyns A, Alexopoulos EI, Ersu R, Joosten K, Larramona H, Miano S, Narang I, Trang H, Tsaoussoglou M, Vandenbussche N, Villa MP, Van Waardenburg D, Weber S, Verhulst S. Obstructive sleep disordered breathing in 2- to 18-year-old children: diagnosis and management. Eur Respir J. 2016 Jan;47(1):69-94. doi: 10.1183/13993003.00385-2015. Epub 2015 Nov 5. PMID 26541535
- [Background] De Luca Canto G, Pacheco-Pereira C, Aydinoz S, Bhattacharjee R, Tan HL, Kheirandish-Gozal L, Flores-Mir C, Gozal D. Adenotonsillectomy Complications: A Meta-analysis. Pediatrics. 2015 Oct;136(4):702-18. doi: 10.1542/peds.2015-1283. Epub 2015 Sep 21. PMID 26391937
- [Background] Kang KT, Hsu WC. Adenotonsillectomy outcomes in treatment of obstructive sleep apnea in children: a multicenter retrospective study. Am J Respir Crit Care Med. 2012 Nov 1;186(9):927; author reply 927-8. doi: 10.1164/ajrccm.186.9.927. No abstract available. PMID 23118085
- [Background] Castorena-Maldonado A, Torre-Bouscoulet L, Meza-Vargas S, Vazquez-Garcia JC, Lopez-Escarcega E, Perez-Padilla R. Preoperative continuous positive airway pressure compliance in children with obstructive sleep apnea syndrome: assessed by a simplified approach. Int J Pediatr Otorhinolaryngol. 2008 Dec;72(12):1795-800. doi: 10.1016/j.ijporl.2008.08.016. Epub 2008 Oct 4. PMID 18835648
- [Background] Monahan KJ, Larkin EK, Rosen CL, Graham G, Redline S. Utility of noninvasive pharyngometry in epidemiologic studies of childhood sleep-disordered breathing. Am J Respir Crit Care Med. 2002 Jun 1;165(11):1499-503. doi: 10.1164/rccm.200111-061OC. PMID 12045123
- [Background] Corda L, Redolfi S, Montemurro LT, La Piana GE, Bertella E, Tantucci C. Short- and long-term effects of CPAP on upper airway anatomy and collapsibility in OSAH. Sleep Breath. 2009 May;13(2):187-93. doi: 10.1007/s11325-008-0219-1. Epub 2008 Sep 25. PMID 18815823